CLINICAL TRIAL: NCT02389361
Title: ZIH Study : Comparison of Oral Zaldiar (Combination of Paracetamol and Tramadol) With Intravenous Paracetamol and Tramadol for Postoperative Analgesia After Inguinal Hernia Repair
Brief Title: Comparison of Oral Zaldiar With Intravenous Paracetamol and Tramadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, Eric DEFLANDRE, MD, FCCP, Astes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASTES - ZIH
Record Dates: First submitted 2015-02-27; First posted 2015-03-17 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Tramadol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Z (Experimental): Postoperative Analgesia with Zaldiar
  Interventions: Drug: Zaldiar
- Group PT (Active Comparator): Postoperative Analgesia with Paracetamol-Tramadol
  Interventions: Drug: Paracetamol-Tramadol

INTERVENTIONS:
Drug: Zaldiar — Postoperative analgesia with oral Zaldiar (combination of tramadol and paracetamol)
  Other Names: Oral Zaldiar
  Arms: Group Z
Drug: Paracetamol-Tramadol — Postoperative analgesia with intravenous Paracetamol and Tramadol
  Other Names: Intravenous Paracetamol and Tramadol
  Arms: Group PT

SUMMARY:
Comparison of two different regimens of analgesia after inguinal hernia repair. First, is a classical intravenous protocol with paracetamol and tramadol. Second is an oral protocol with Zaldiar (combination of paracetamol and tramadol).

DETAILED DESCRIPTION:
Comparison of two different regimens of analgesia after inguinal hernia repair. First, is a classical intravenous protocol with paracetamol and tramadol. This is the classical approach. Second is an oral protocol with Zaldiar (combination of paracetamol and tramadol). This is the new approach.

ELIGIBILITY:
Inclusion Criteria:

* All patients incoming for inguinal hernia repair

Exclusion Criteria:

* Preoperative abuse of analgesics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, Study Director — Astes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Z | Group PT
Started | 24 | 27
Completed | 24 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Z | Group PT | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 20 | 34
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.08 (16.42) | 62.41 (14.51) | 57.19 (15.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 21 | 24 | 45
Region of Enrollment [Number; unit: participants]
  Belgium | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Acute Pain
Description: Difference between groups in term of analgesia (as measured by Visual Analog Scale: VAS). The VAS range are between 0 and 10. A worse outcome was defined as VAS > 4. The VAS use units on a scale.
Time Frame: In recovery room
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Group Z | Group PT
Number analyzed (Participants) | 24 | 27
units on a scale | 1.5 (1.28) | 1.74 (1.86)

ADVERSE EVENTS:
Arm/Group | Group Z | Group PT
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No